CLINICAL TRIAL: NCT04691869
Title: Quantitative Ultrasound Use to Increase Geriatric Follow-up for Osteoporosis
Acronym: QUS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We were not able to complete the study due to COVID restrictions and never enrolled any participants.
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Carol A. Lin, MD, Associate Residency Program Director, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: STUDY00000291
Record Dates: First submitted 2020-12-09; First posted 2020-12-31 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Osteoporosis; Bone Loss
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control (No Intervention): Patients will be randomized into a control group and study group. The control group will receive an informational discussion with the nurse-practitioner regarding steps to reduce the risk for osteoporosis, as well as an informational handout in their discharge papers.
- Interventional (Experimental): The study group will undergo the QUS (performed by a member of the study team) and receive the same informational discussion and handouts, with the addition of a QUS screening to take to their follow-up appointment. The QUS screening will come with a half-page description, describing the screening and what their results mean. A discussion lead by the nurse-practitioner, who is a member of the study staff, regarding the results will happen prior to discharge.
  Interventions: Device: Achilles EXPII

INTERVENTIONS:
Device: Achilles EXPII — Portable ultrasound machine that measures a patient's bone density at the calcaneus.
  Arms: Interventional

SUMMARY:
The objective of this study is to determine whether patient follow up for osteoporosis is aided using a quantitative ultrasound (QUS) measurement.

Using the QUS measurement could potentially improve osteoporosis follow-up rates, and in-office patient measurements have been previously shown to increase compliance with treatment in other conditions. Increased compliance with follow-ups and medication recommendations have been shown to decrease fracture rates in patients with osteoporosis.

DETAILED DESCRIPTION:
Over 10 million Americans have osteoporosis, which is defined as a chronic, progressive disease presenting with deterioration of bone tissue and fragility subsequently leading to an increased fracture risk1. A positive diagnosis for osteoporosis is significantly correlated with increased age, making geriatrics patients an at-risk group for bone health complications2. A pathophysiological diagnosis for osteoporosis is done radiographically based on bone mineral density from a dual energy x-ray absorptiometry assessment (DXA)3. DXA scans have been used increasingly over time in geriatric populations to screen patients for osteoporosis4; however, one problem with DXA scans is the radiation dose due to x-ray radiography4. Therefore, using DXA scans as a preliminary screening method comes with risks, even though it is the gold standard for diagnosis3.

Osteoporosis is often referred to as a silent disease because people are not aware that they have low bone density9. The first sign may be loss of height but can also be a fracture due to a ground level mechanical fall. As people age, their bones lose their strength (density) and become more brittle2,10. Unfortunately, fractures can have devastating effects on people's quality of life causing chronic pain, difficulties with mobility, need for increased assistance, isolation, increased nursing home placement and rates of death10. Also, once a person has fallen and had a fragility fracture, they are likely to do so again10. Our goal is to encourage older adult patients to follow-up with their doctors to discuss osteoporosis screening, diagnosis, and treatment to help reduce the prevalence of fragility fractures.

Osteoporosis follow-up rates need to be improved in geriatric populations. Increased compliance with follow-ups and medication recommendations have been shown to decrease fracture rates in this population5. In-office patient measurements have been previously shown to increase compliance with treatment. In the case of smoking, carbon monoxide (CO) monitors increased a patient's willingness to comply with cessation protocols significantly in an orthopedic fracture population6.

Quantitative ultrasound scans (QUS) have emerged as a simple point-of-care test for bone density. 7 For a quantitative ultrasound scan, the patient sits in a chair and places their heel on specialized ultrasound machine in a manner similar to having the size of the foot measured at a department store. The machine is portable and can be performed at the bedside. Prior research has demonstrated that, although QUS cannot replace DXA scans as the gold standard for diagnosis of osteopenia, it can still be used to immediately identify abnormal bone density8. Integrating QUS scans into geriatric fracture treatment comes at little risk, and, similar to home CO monitoring for smoking cessation, may provide additional information to the patient to encourage further action.

ELIGIBILITY:
Inclusion Criteria:

* At least 65 years of age (DXA scan is not covered until 65 years of age)
* Presents with pelvic or extremity fracture(s) to the hospital

Exclusion Criteria:

* Previous diagnosis of osteoporosis with active treatment
* Multi-system injury patients (eg: brain, thoracic, spine, and intrabdominal)
* Patients with a pre-existing condition of advanced dementia
* Patients who lack the capacity to consent
* If a patient is unable to consent in English

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Osteoporosis Care | Up to 3 months after patient enrollment in study
  Percent of patients who follow-up within 3 months with a primary care physician, geriatrician, rheumatologist or an endocrinologist to discuss osteoporosis care.

SECONDARY OUTCOMES:
DXA Scan within 6 months after patient follows-up with physician, geriatrician, rheumatologist or an endocrinologist | Up to 6 months after patient follow up in study
  Percent of patients who follow-up within 6 months receive a DXA scan.
Percent of patients prescribed pharmacological therapy for bone health treatment who received a DXA scan and were diagnosed with osteoporosis | At the time of DXA scan
  For patients who received a DXA scan and were then diagnosed with osteoporosis, what percent of patients those were prescribed pharmacological treatment for bone health.

CONTACTS AND LOCATIONS:
Overall Officials: Carol Lin, MD, Principal Investigator — Cedars-Sinai Medical Center